CLINICAL TRIAL: NCT02755038
Title: Scalp Hair Estradiol and Progesterone Level Determination in Pre-menopausal and Post-menopausal Women (Proof of Concept Study)
Brief Title: Scalp Hair Estradiol and Progesterone Level Determination in Women (Proof of Concept Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, samer.khoury, Dr, Bnai Zion Medical Center
Other Study IDs: BNZ160015CTIL
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: postmenopausal women; scalp hair; estrogen; progesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Scalp Hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- premenopausal and postmenopausal women: One group will include 20 premenopausal women under the age 40 years old, with regular menstruation cycles and without any illness or medication including birth control pills or steroidal ointments, and without known diagnosis of polycystic ovaries or fertility disorder. The second group will include 20 postmenopausal women over the age of 60, with no menstruation at least for the last five years, and without hormone therapy or treatment of any Steroidal therapy for the last year.

SUMMARY:
The investigators hypothesis is that we can determine estrogen and progesterone levels in the hair by using the immune method and we can show a significant difference in the levels of these hormones in both groups of women: pre- and postmenopausal women. If indeed it would then be possible in future to carry out research that can find a relationship between the levels of these hormones and various diseases

DETAILED DESCRIPTION:
One group will include 20 women under the age 40 years old, with regular menstruation cycles and without any illness or medication including birth control pills or steroidal ointments, and without known diagnosis of polycystic ovaries or fertility disorder. The second group will include 20 women over the age of 60, with no menstruation at least for the last five years, and without hormone therapy or treatment of any Steroidal therapy for the last year.

From all of the participants the investigators will collect hair samples at the crown back of the head (hair will be cut as close as possible to the scalp), the samples will be measured quantitatively about 100 hairs at a length of 2-3 cm. In order to grind the hair samples we will use a mini-Bead beater machine. milled hairs will be incubated overnight in a solution of 1 ml methanol 50, in constant gentle muddling. Afterwards, ethanol will disperse through a stream of nitrogen. The remainder of the suspension will be dissolved at 200 microliter buffer PBS (Phosphate-Buffered Saline) (pH 8.0) and the concentration of estrogen and progesterone will be measured by using the immune method which is available in the endocrine laboratory in Bnai Zion medical center. At the end of the study the investigators will cary out a statistical comparison of progesterone and estrogen levels between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* women under 40 with regular cycles
* Women over the age of 60 in menopause for at least 5 years

Exclusion Criteria:

* pregnant women
* oral contraceptive treatment in the last year
* hormonal replacement therapy in the last year
* 6 month after delivery
* infertile women
* irregular menstruation
* women with progesterone secretion intrauterine device in the last year
* BMI- Body Mass Index- below 25 or above 35
* Polycystic Ovarian Syndrome
* steriodal treatment including inhalers and ointments.
* status post Removal of the ovaries or uterus
* Breast or uterine cancer in the past.
* any pituitary or adrenal disease

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One group will include 20 women under the age 40 years old, with regular menstruation cycles and without any illness or medication including birth control pills or steroidal ointments, and without known diagnosis of polycystic ovaries or fertility disorder. The second group will include 20 women over the age of 60, with no menstruation at least for the last five years, and without hormone therapy or treatment of any Steroidal therapy for the last year.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
concentration of hair scalp progesterone | 3 months
  concentration of hair scalp progesterone (nmol\L)
concentration of hair scalp estrogen | 3 months
  concentration of hair scalp estrogen (pmol\L)

CONTACTS AND LOCATIONS:
Overall Officials: samer khoury, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Samer Khoury, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No